CLINICAL TRIAL: NCT05927415
Title: A Phase 1, Open-label, Study to Evaluate the Pharmacokinetics of Efgartigimod IV 10 mg/kg Single Dose Administered in Participants With Renal Impairment
Brief Title: A Study to Test How Kidney Problems Influence the Blood Concentrations of Efgartigimod
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ARGX-113-2201
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mild renal impairment (Experimental): Patients with 60 <= eGFR <90
  Interventions: Biological: Efgartigimod IV
- Moderate renal impairment (Experimental): Patients with 30 <= eGFR <60
  Interventions: Biological: Efgartigimod IV
- Severe renal impairment (Experimental): Patients with eGFR <30
  Interventions: Biological: Efgartigimod IV
- Normal renal function (Experimental): Patients with eGFR >=90
  Interventions: Biological: Efgartigimod IV

INTERVENTIONS:
Biological: Efgartigimod IV — Intravenous infusion of efgartigimod

SUMMARY:
A study to test how kidney problems influence the blood concentrations of efgartigimod

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 and ≤80 years of age when signing the informed consent form, and willing and able to understand and comply with the requirements of the study
* Participant has BMI ≥18.0 and ≤38.0 kg/m2
* Female participant of childbearing potential agrees to contraceptive use consistent with local regulations for clinical studies and has a negative serum pregnancy test
* Participant has a stable diagnosis of RI, without any significant change in overall disease status in the 3 months before screening
* At screening, the participant has eGFR (mL/min) calculated using the CKD-EPI equation that is within the following ranges: 60 to <90 (mild RI); 30 to <60 (moderate RI); <30 (severe RI not requiring dialysis); ≥90 (normal renal function)
* Participant has normal or not clinically significant findings in physical examination, vital signs, ECG, and clinical laboratory evaluations; exceptions may be granted for findings consistent with the participant's RI or other related stable diseases
* Absence of clinically significant illness and surgery during the 4 weeks before the infusion and absence of clinically significant history of hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, and immunologic disease
* Participant with RI is receiving a stable medical regimen for 14 days before the efgartigimod infusion, except for routine daily management of electrolytes (eg, potassium), acid-base, or other electrolyte abnormalities associated with RI. Control participant agrees to not receive any medications, except contraceptives and occasional paracetamol use

Exclusion Criteria:

* Participant has previously participated in an efgartigimod clinical study and received at least 1 dose
* Participant has a known hypersensitivity to 1 of the components in efgartigimod IV or a history of severe allergic or anaphylactic reactions
* Participant has a condition except for RI that could affect efgartigimod PK
* Participant has a clinically significant unstable medical condition or history of any illness that can increase the risk associated with study participation or efgartigimod administration or can interfere with the interpretation of study results and make the participant inappropriate for this study.
* Participant has a positive nasopharyngeal swab test for SARS-CoV-2 on day -1
* Participant has supine 12-lead ECG abnormalities at screening considered clinically significant and clinically significant vital sign abnormalities
* Participant has a history of significant drug or alcohol abuse within 6 months before screening, or positive urine drug screen or alcohol test at screening
* Participant has a history of malignancy unless considered to be cured by adequate treatment with no evidence of recurrence for ≥3 years before the efgartigimod infusion. Participants with the following cancers can be included at any time, provided they are adequately treated before they participate in the study: Basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Incidental histological finding of prostate cancer
* Participant has a clinically significant active or chronic, bacterial, viral, or fungal infection at screening, including a positive serum test at screening for active infection with any of the following conditions: HBV indicative of an acute or chronic infection unless associated with a negative HBsAg or negative HBV DNA test, HCV based on HCV antibody assay unless an RNA test indicates the participant is HCV negative, HIV based on CD4 count <200 cells/mm3 associated with an AIDS-defining condition, HIV based on CD4 count greater than 200 cells/mm3 not adequately treated with antiretroviral therapy
* Participant has participated in a clinical study involving the administration of an IMP or marketed drug or device within 30 days of the infusion, administration of a biological product in the context of a clinical study within 90 days of the infusion, or concurrent participation in an investigational study involving no drug or device administration
* Participant is an employee of the investigator or study site with direct involvement in this clinical study or other studies under the direction of the investigator or study site or a family member of an employee of the investigator
* Female participant has a positive pregnancy test before dosing or is pregnant or breastfeeding
* Participant has had a renal transplant
* Participant has received any new prescription medication before the efgartigimod infusion or other medication, except those approved by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Efgartigimod PK parameters (Cmax) | up to 64 days

SECONDARY OUTCOMES:
Efgartigimod urine concentrations | up to 64 days
Incidence of serious adverse events | up to 64 days
Reduction from baseline in total IgG levels over time | up to 64 days
Incidence of ADA to efgartigimod | up to 64 days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel GmbH, Kiel
  - APEX GmbH, Munich